CLINICAL TRIAL: NCT03595371
Title: A Pilot, Open-Label, Phase 2, Single-Center, Repeat Dose, Proof- Of-Concept Safety, Pharmacodynamics and Efficacy Study of Orally Administered Dapansutrile Capsules in Subjects With Schnitzler's Syndrome
Brief Title: Pilot Study of Dapansutrile Capsules in Schnitzler's Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to study design issues that did not allow for determination of efficacy and safety in subjects with Schnitzler Syndrome who are currently well controlled on anakinra therapy.
Sponsor: Olatec Therapeutics LLC (Industry)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OLT1177-07
Record Dates: First submitted 2018-06-11; First posted 2018-07-23 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-01

CONDITIONS: Schnitzler Syndrome
Keywords: Schnitzler
MeSH Terms: conditions — Schnitzler Syndrome | interventions — dapansutrile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- dapansutrile capsules (Experimental): Hard gelatin capsules containing 100 mg of dapansutrile (API)
  Interventions: Drug: dapansutrile

INTERVENTIONS:
Drug: dapansutrile — 500 mg dapansutrile administered twice daily (with a potential to increase the dosage to 2 g dapansutrile daily) for a duration of up to 14 consecutive days.
  Other Names: OLT1177 capsules

SUMMARY:
This is a pilot, open-label Phase 2, single-center, repeat dose, single cohort, proof-of-concept, safety, pharmacodynamics and efficacy study of dapansutrile capsules to be conducted in subjects with Schnitzler's syndrome (SchS) currently well controlled by anakinra therapy. At least 5 but no more than 10 subjects will be enrolled.

DETAILED DESCRIPTION:
Subjects who are currently taking and responsive to anakinra (Kineret®) for at least 6 weeks will be screened for eligibility at the Screening / Baseline (Day 1) visit. Following confirmation of eligibility, subjects will be enrolled, the first dose of dapansutrile will be administered at the clinical site and safety and efficacy assessments will be completed. Subjects will self-administer dapansutrile twice a day by mouth for 14 consecutive days. Subjects will continue their standard dose of anakinra for Days 1, 2 and 3 of the 14-day Treatment Period and will then cease taking anakinra. At the end of the 14-day Treatment Period subjects will remain off all medication for Schnitzler's syndrome and at the first signs of a relapse or worsening of SchS symptoms, subjects will visit the study clinic for the Symptom Onset visit (SOV) to determine with the Investigator when injections of anakinra should be resumed. In addition, subjects will return to the study clinic on Days 5, 9, 14, 15,16, 18 and 21 for follow-up visits1 and will be contacted by telephone on Day 42 (± 3 Days) for additional follow-up. The Day 15 (± 1 day), Day 16 (± 1 day) and Day 18 (± 1 day) visits will only occur if anakinra therapy has not yet been resumed.

Subjects will be given the option to remain in the Nijmegen area after the Day 14 visit and return to the study clinic for the Day 15, 16 and 18 follow-up visits. Alternatively, subjects will be given the option to have these visits conducted at their home by a trained study nurse.

Safety assessments will be conducted at each visit and subjects will capture the frequency and intensity of symptoms, including body temperature, using a paper diary. Safety and tolerability will be evaluated by monitoring the occurrence of adverse events (AEs) and changes in abbreviated physical examination findings, vital signs and clinical safety laboratory test results (chemistry, hematology and urinalysis) and inflammatory biomarkers. Clinical activity will be evaluated by: Subject Diary (completed daily), Subject Global Assessment of Disease Activity, Investigator Global Assessment of Disease Activity, and analysis of biomarkers of inflammation, including changes in C-reactive protein (CRP). Daily diary assessments will be captured starting at the Screening / Baseline (Day 1) visit and will continue until Symptom Onset visit or Day 21 visit (whichever occurs latest).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 18 years old or older
2. Prior diagnosis of Schnitzler's syndrome
3. Presence of Schnitzler's syndrome that is well controlled by and responsive to anakinra for at least 6 weeks prior to the Screening/Baseline visit
4. Grade 0 SchS symptoms at the Screening/Baseline visit
5. Acceptable overall medical condition to be safely enrolled in and to complete the study (with specific regard to cardiovascular, renal and hepatic conditions) in the opinion of the Investigator
6. Ability to provide written informed consent prior to initiation of any study-related procedures, and ability, in the opinion of the Investigator, to understand and comply with all the requirements of the study as outlined in the protocol.

Exclusion Criteria:

1. Pregnant, nursing or intent to become pregnant during the study
2. Not responsive or well controlled by anakinra therapy for at least 6 weeks prior to the Screening/Baseline visit
3. Use or planned use of any prohibited concomitant medications/therapies such as immunotherapies or corticosteroids during the study (until relapse and resumption of anakinra injections)
4. Active infection within 3 days prior to the Screening/Baseline visit
5. History of or known positive for HIV, Hepatitis B surface antigen (HBsAg) or antibodies to Hepatitis C Virus (HCV)
6. Any other concomitant medical or psychiatric conditions, including alcohol or substance abuse, diseases or prior surgeries that in the opinion of the Investigator would impair the subject from safely participating in the trial and/or completing protocol requirements
7. Enrollment in any trial and/or use of any investigational product or device within the immediate 30-day period prior to the Screening/Baseline visit
8. Enrollment in any study previously sponsored by Olatec Therapeutics LLC, specifically Study OLT1177-01, Study OLT1177-02, Study OLT1177-03, Study OLT1177-04 or Study OLT1177-05

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
Schnitzler's Syndrome Symptom Index | Day 14
  Proportion of subjects with Grade 0 or 1 SchS symptoms at end of treatment. The Schnitzler's Syndrome Symptom Index (SchS Index) is a composite index incorporating the investigator global assessment of disease activity and levels of plasma CRP. The SchS Index is graded on a 0 - 3 scale with 0 being the best score and indicating "no symptoms of Schnitzler's syndrome" and 3 being the worst score and indicating "severe symptoms of Schnitzler's syndrome".

SECONDARY OUTCOMES:
Physical Examination | Day 14
  A full or targeted physical examination of the patient's major body systems
Vital signs - pulse | Day 14
  Pulse will be recorded and analyzed for changes.
Vital signs - temperature | Day 14
  Body temperature will be recorded and analyzed for changes.
Vital signs - respirations | Day 14
  Respiration rate will be recorded and analyzed for changes.
Vital signs - blood pressure | Day 14
  Systolic and diastolic blood pressure will be recorded and analyzed for changes.
Safety laboratory measures - chemistry markers | Day 14
  Blood samples will be drawn and analyzed for chemistry blood markers.
Safety laboratory measures - hematology/complete blood count | Day 14
  Blood samples will be drawn and a complete blood count will be performed.
Safety laboratory measures - urinalysis | Day 14
  Urine samples will be collected and analyzed.
Adverse events | Up to 42 days
  Adverse events will be described with respect to seriousness, intensity, relationship to treatment, action taken and outcome of the event.
Photographs of posterior torso | Day 14
  Photographs of posterior torso or other non-identifying areas of the body displaying urticarial rash.
Investigator Global Assessment of Disease Activity | Later of Day 14 or symptom relapse (expected no later than Day 28)
  One general question the Investigator is asked to answer about the overall perceived status of the subject's symptoms.
Subject Global Assessment of Disease Activity | Later of Day 14 or symptom relapse (expected no later than Day 28)
  Overall assessment of disease activity in response to the question: Please note on this scale (0=bad; 10=outstanding) how you are feeling.
Subject Skin Assessment | Later of Day 14 or symptom relapse (expected no later than Day 28)
  Extent of urticaria on subject's body.
Time to relapse of SchS Symptoms after cessation of dapansutrile | Later of Day 14 or symptom relapse (expected no later than Day 28)
  Time to the emergence of Grade 2 or higher SchS symptoms
Subject Global Evaluation of Treatment | Later of Day 14 or symptom relapse (expected no later than Day 28)
  Two general questions the subject is asked to answer about the overall perceived quality of the investigational product.

OTHER OUTCOMES:
Plasma concentrations of dapansutrile | Later of Day 14 or symptom relapse (expected no later than Day 28)
  Blood samples analyzed for levels of dapansutrile.

CONTACTS AND LOCATIONS:
Overall Officials: Curt Scribner, MD, Study Chair — Olatec Therapeutics LLC
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No